CLINICAL TRIAL: NCT01766284
Title: Study of the Diagnostic Efficacy of "Real Time" Niris 1300e Optical Coherence Tomography (OCT) Imaging System in the Management of Pre-invasive and Invasive Neoplasia of the Uterine Cervix (PUSHOCTII)
Brief Title: Study of the Diagnostic Efficacy of "Real Time" Niris 1300e Optical Coherence Tomography (OCT) Imaging System in the Management of Pre-invasive and Invasive Neoplasia of the Uterine Cervix
Acronym: PUSHOCTII
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Preventive Oncology International, Inc. (Other)
Collaborators: Imalux (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PUSHOCTII
Record Dates: First submitted 2012-11-04; First posted 2013-01-11 (Estimated); Last update posted 2013-02-15 (Estimated); Status verified 2013-02

CONDITIONS: Cervical Intraepithelial Neoplasia; Cervix Cancer; Cervical Dysplasia; CIN; Human Papillomavirus
Keywords: Human Papillomavirus; Optical Coherence Tomography; Imaging Systems; Cervical intraepithelial neoplasia; Cervical Cancer; Cervical Dysplasia
MeSH Terms: conditions — Uterine Cervical Dysplasia; Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Niris 1300e OCT imaging (Experimental): OCT imaging of the cervix using Niris 1300e will include computer aided calculations for epithelial brightness.
  Interventions: Device: NIRIS 1300e

INTERVENTIONS:
Device: NIRIS 1300e — Optical coherence tomography (OCT) is similar to ultrasound pulse-echo imaging, with optical scatter rather than acoustic reflectivity being measured. OCT employs harmless near-infrared light technology which uses low coherence interferometry to produce an image (based on optical scattering) of tissue microstructure.

SUMMARY:
Optical Coherence Tomography (OCT) is a technology using harmless near infra-red light scatter to produce an image. Prior studies with OCT have demonstrated that OCT of the uterine cervix can differentiate between grades of pre-invasive and invasive cervical disease and cancer. This study will evaluate the ability of the NIRIS 1300e imaging (OCT) system to detect pre-invasive cervical disease and cervical cancer.

DETAILED DESCRIPTION:
B. Specific Aims

1. Primary. To determine the sensitivity, specificity, positive and negative predictive values for Niris 1300e OCT enhanced gynecologic examination (VIA-OCT vs.colposcopy-biopsy) for the detection of lesions equal or greater than cervical intraepithelial neoplasia II (CIN II) and cancer in a "real time" clinical evaluation.
2. Secondary. To examine the ease of use of Niris 1300e OCT in a real time clinical setting in order to assess its potential application during a "see and treat" or "single episode of care" clinic visit.

ELIGIBILITY:
Inclusion Criteria:

1. Female subjects > 18 years of age
2. Subject must voluntarily sign a Patient Informed Consent Form specific to the study.
3. Subject must be physically and mentally willing to comply with all study requirements, especially conduct of a colposcopy exam.
4. Participant must be attending the Center for Cervical Diagnosis.

Exclusion Criteria:

1. Based on clinical history, physical exam and patient presentation, the subject is unable to provide adequate informed consent and/or comply with the study requirements.
2. Subject is a prisoner.
3. Subject is pregnant.
4. Subject has had a hysterectomy
5. Subject has received prior pelvic radiotherapy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2012-11; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
To determine the accuracy of VIA plus Niris 1300e OCT enhanced gynecologic examination. | Study will be completed over a 4 day period with OCT and brightness determination as each patient is seen. During the next 4 months, we will conduct blinded reviews of the images to determine new sets of brightness numbers.

SECONDARY OUTCOMES:
To compare OCT image (Niris 1300e) technology directly to colposcopy with biopsy for the detection of lesions equal or greater than cervical intraepithelial neoplasia II (CIN II) and cancer in a "real time" clinical evaluation. | Study will be completed over a 4 day period with OCT and brightness determination as each patient is seen. During the next 4 months we will conduct blinded reviews of the images to determine new sets of brightness numbers.

CONTACTS AND LOCATIONS:
Overall Officials: Jerome L Belinson, MD, Principal Investigator — Preventive Oncology International; Rufiang Wu, MD, Principal Investigator — Peking University Shenzhen Hospital
Locations (1):
- Peking University Shenzhen Hospital, Shenzhen, Guangdong, China

REFERENCES:
- [Background] Wulan N, Rasool N, Belinson SE, Wang C, Rong X, Zhang W, Zhu Y, Yang B, Tresser NJ, Mohr M, Wu R, Belinson JL. Study of the diagnostic efficacy of real-time optical coherence tomography as an adjunct to unaided visual inspection with acetic acid for the diagnosis of preinvasive and invasive neoplasia of the uterine cervix. Int J Gynecol Cancer. 2010 Apr;20(3):422-7. doi: 10.1111/IGC.0b013e3181d09fbb. PMID 20375808
- [Background] Liu Z, Belinson SE, Li J, Yang B, Wulan N, Tresser NJ, Wang C, Mohr M, Zhang L, Zhou Y, Weng L, Wu R, Belinson JL. Diagnostic efficacy of real-time optical coherence tomography in the management of preinvasive and invasive neoplasia of the uterine cervix. Int J Gynecol Cancer. 2010 Feb;20(2):283-7. doi: 10.1111/IGC.0b013e3181cd1810. PMID 20134271
- [Background] Belinson SE, Ledford K, Rasool N, Rollins A, Wilan N, Wang C, Rong X, Zhang W, Zhu Y, Tresser N, Wu R, Belinson JL. Cervical epithelial brightness by optical coherence tomography can determine histological grades of cervical neoplasia. J Low Genit Tract Dis. 2013 Apr;17(2):160-6. doi: 10.1097/LGT.0b013e31825d7bf0. PMID 23343696
- See also: Preventive Oncology International, Inc. — http://www.poiinc.org